CLINICAL TRIAL: NCT03580460
Title: Cultural Adaptation and Piloting of an Avatar Delivered Smoking Cessation Intervention for Low Income Smokers in Baltimore City Living With HIV
Brief Title: Cultural Adaptation and Piloting of a Smoking Cessation Intervention for Smokers With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00117151
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hiv; Cigarette Smoking
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: 2 arm, RCT with waitlist control
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (No Intervention): After 8 weeks, individuals randomized to this arm receives the computer-delivered smoking cessation counseling intervention
- Computer Delivered Intervention (Experimental): Individuals receive a 15-20 minute computer delivered smoking cessation counseling intervention
  Interventions: Behavioral: Computer delivered smoking cessation counseling

INTERVENTIONS:
Behavioral: Computer delivered smoking cessation counseling — 15 to 20 minute computer-delivered interactive smoking cessation counseling
  Arms: Computer Delivered Intervention

SUMMARY:
One population of tobacco users that is severely affected by the consequences of smoking is people living with HIV (PLWH). Between 40-84% of PLWH smoke, a percentage that has remained constant since the first studies of smoking in HIV were conducted in the 1990's. Overall, smoking related morbidity and mortality is also greatly increased among PLWH smokers. Compared with PLWH nonsmokers, PLWH who smoke have more than 5 times the risk of non-HIV-related mortality and almost 4 times the risk of all-cause mortality. Compared with the general population, incidence ratio of smoking related cancers (eg, lung, head, neck, bladder and esophageal) is more than 5 times higher. At a critical time when advances in HIV care are providing an opportunity for prolonged life, smoking is significantly impeding the health of PLWH.

To produce meaningful changes in smoking, however, treatment will have to be acceptable and engaging to this population as well as feasible and sustainable to implement in a busy clinic. Novel technology-based interventions that incorporate evidence-based behavioral and pharmacologic interventions for smoking and are culturally tailored offer real solutions to these implementation barriers. Research shows that internet- or computer-delivered interventions (CDI) that are tailored and interactive can be efficacious in reducing smoking and are significantly more effective than usual care or written self-help materials. CDIs can also be readily adapted to different sociodemographic characteristics of a patient population because content is modular and menu driven. Moreover, technology-based interventions appear as effective as counselor-delivered interventions in reducing smoking. This growing body of evidence strongly suggests that these interventions offer promise in reducing smoking, the potential to reach significantly more patients, and the ability to overcome barriers of cost, implementation, and cultural nonspecificity. The goal of this pilot study is test to examine feasibility, acceptability of a computer-delivered smoking cessation intervention for PLWH, and to determine if intervention participation results in increased readiness to quit smoking and increased confidence in ability to quit smoking.

DETAILED DESCRIPTION:
One population of tobacco users that is severely affected by the consequences of smoking is people living with HIV (PLWH). Between 40-84% of PLWH smoke, a percentage that has remained constant since the first studies of smoking in HIV were conducted in the 1990's. Overall, smoking related morbidity and mortality is also greatly increased among PLWH smokers. Compared with PLWH nonsmokers, PLWH who smoke have more than 5 times the risk of non-HIV-related mortality and almost 4 times the risk of all-cause mortality. Compared with the general population, their incidence ratio of smoking related cancers (eg, lung, head, neck, bladder and esophageal) is more than 5 times higher. At a critical time when advances in HIV care are providing an opportunity for prolonged life, smoking is significantly impeding the health of PLWH.

To produce meaningful changes in smoking, however, treatment will have to be acceptable and engaging to this population as well as feasible and sustainable to implement in a busy clinic. Novel technology-based interventions that incorporate evidence-based behavioral and pharmacologic interventions for smoking and are culturally tailored offer real solutions to these implementation barriers. Research shows that internet- or computer-delivered interventions (CDI) that are tailored and interactive can be efficacious in reducing smoking and are significantly more effective than usual care or written self-help materials. CDIs can also be readily adapted to different sociodemographic characteristics of a patient population because content is modular and menu driven. Moreover, technology-based interventions appear as effective as counselor-delivered interventions in reducing smoking. This growing body of evidence strongly suggests that these interventions offer promise in reducing smoking, the potential to reach significantly more patients, and the ability to overcome barriers of cost, implementation, and cultural nonspecificity. The goal of this pilot randomized controlled trial (RCT) is study is test to examine feasibility, acceptability of a computer-delivered smoking cessation intervention for PLWH, and to determine if intervention participation results in increased readiness to quit smoking and increased confidence in ability to quit smoking.To pilot test the computer-delivered intervention among 40 individuals with HIV receiving care in an urban HIV clinic in a small Randomized Controlled Trial 2a) To determine intervention effect on 1) readiness to quit smoking 2) increased confidence in ability to quit smoking 2) uptake of smoking cessation therapy, including a. Quit Line, b. Nicotine replacement therapy c. Pharmacotherapy (varenicline, Wellbutrin) Hypothesis: Investigators hypothesize that intervention participation will be associated with 1) increased readiness to quit and confidence in quitting smoking and 2) increased engagement with smoking cessation services.

2b) To examine feasibility and acceptability of delivering the computer-delivered smoking cessation counseling in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* A patient in the Johns Hopkins University (JHU) Bartlett Clinic
* Smoked >100 cigarettes in their lifetime
* Current daily smoker (verified by exhaled carbon monoxide)
* English speaking.

Exclusion Criteria:

* Individuals will be excluded if they do not meet the above requirements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Readiness to change smoking behaviour | immediately post-intervention
  Self-report on the Alcohol and Other Drug Contemplation Ladder, 1-10 Visual Analog Scale with 0- no readiness and 10- full readiness

SECONDARY OUTCOMES:
Engagement in Smoking Cessation Services | 8 weeks post-intervention
  Self-Reported Use of Quitline or pharmacotherapy for smoking cessation which will based on a questionnaire.
Confidence in ability to quit smoking | immediately post-intervention
  Self report on visual analog scale measuring confidence in ability to quit smoking on visual analog scale 1-100 with a higher value representing higher confidence

CONTACTS AND LOCATIONS:
Overall Officials: Geetanjali Chander, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States